CLINICAL TRIAL: NCT03755284
Title: The Effect Of Sacral Massage On Labour Pain and Anxiety: A Randomized Controlled Trial
Brief Title: The Effect of Sacral Massage on Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semra Çevik, phD (Other)
Responsible Party: Sponsor-Investigator, Semra Çevik, phD, Assiatant Professor, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sacral Massage
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Labor Pain
Keywords: anxiety; labor pain; massage; surveys and questionnaires; visual analog scale
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized and controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacral Massage Group (Experimental): The massage was applied only to the pregnant women in the intervention group at every phase of labour. There was no intervention in the control group except for routine hospital applications. The steps taken in this study are discussed below.
  For the pregnant women included in the experimental group:
  In addition to providing them with routine nursing/midwifery care, the women in the experimental group were administered a massage to the sacral region under the supervision of a doctor for 30 minutes using the effleurage (patting) ( 15 minutes) and vibration technique ( 15 minutes) in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour. To achieve this, the patients were placed in the left lateral position in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour.
  Interventions: Other: Sacral Massage
- Control Group (No Intervention): There was no intervention in the control group except for routine hospital applications. The steps taken in this study are discussed below.
  One-on-one interviews were conducted with the pregnant women, and the voluntary disclosure forms, which explained the purpose of the study, were completed.
  The prepared questionnaire form was applied. Routine nursing/midwifery care was applied. The state-trait anxiety inventory (STAI FORM TX-I) was applied and evaluated in the active (5-7 cm) phase.
  The Visual Analogue Scale (VAS) was evaluated once in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases.
  Birth action follow-up form and postpartum interview forms were applied

INTERVENTIONS:
Other: Sacral Massage — ● In addition to providing them with routine nursing/midwifery care, the women in the experimental group were administered a massage to the sacral region under the supervision of a doctor for 30 minutes using the effleurage (patting) ( 15 minutes) and vibration technique ( 15 minutes) in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour. To achieve this, the patients were placed in the left lateral position in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour.
  Arms: sacral Massage Group

SUMMARY:
Nonpharmacologic pain control methods, which are increasingly becoming widespread in coping with the labour pain, are the methods that allow women to completely relax without using any medication and direct them to perceive the pain at the lowest level. This study was conducted to determine the effect of sacral massage, on labour pain and anxiety. This study was conducted as a randomized controlled experimental study at Bağcılar Training and Research Hospital, Obstetrics and Gynecology Clinic between March and October 2016.

Hypotheses of the Study

1. Massage applied to the sacral region decreases the perception of a woman's labour pain.
2. Massage applied to the sacral region decreases the woman's levels of concern and anxiety about labour.
3. Massage applied to the sacral region increases the woman's satisfaction with the labour

DETAILED DESCRIPTION:
Study design

This was a randomized and controlled experimental study aimed to determine the effects of sacral massage on labour pain and anxiety.

Setting and samples

The study was performed in volunteer pregnant women who applied to xxx Training and Research Hospital, Delivery Unit, to undergo their first labour between January 25 and October 25, 2016. This unit contains 1 delivery room (with 2 tables), 2 labour follow-up rooms (with 5 beds), 1 postpartum room (with 5 beds) and 1 nursing room.

According to hospital records, in all, 342 pregnant women who applied to xxx Training and Research Hospital, Delivery Unit to undergo their first labour between January 25 and October 25, 2016, constituted the population of the study. The following inclusion criteria were used to determine participation in the study: (1) 19-40-year-old primiparous pregnant women;(2) Singleton pregnancies between 38-42 weeks; (3) Pregnant women whose labour began spontaneously; (4) Pregnant women with a healthy foetus; (5) Pregnant women without any complications that may cause dystocia during labour; (6) Pregnant women for whom analgesia and anaesthesia were not used during the first phase of labour; (7) Pregnant women who volunteered to participate in the research and who could establish verbal communication. In addition, Pregnant women with high-risk pregnancies, with caesarean section indication, and Pregnant women with a chronic illness were excluded.

The sample size was calculated by Medical Faculty Biostatistics Department using Minitab Program. The sample volume to represent the population was determined as minimum 30 people for each group when considering comparison results of mean scores in the study of Field., with a risk of α= 0.05, an accuracy rate of 1-α =0.95 and a power ratio of B= 0.20, 1-B= 0.80.

The study was conducted with two groups, namely Massage Group (experimental), and Control Group. 30 pregnant women were included in each group; therefore, the study was conducted with a total of 60 pregnant women. The women who participated in the study were randomized randomly as control (double) and experimental (single) groups according to the single or double patient admission numbers. The women who participated in the study were randomized into either the control (double) or the experimental (single) group according to single or double patient admission numbers.

Measurements

In this study, the Questionnaire form, Birth action follow-up form, postpartum interview form ,Visual analogue scale (VAS) and State-trait anxiety inventory (STAI FORM TX-I) were used to collect the data.

1. Questionnaire Form: Questions that reflect the sociodemographic characteristics of the patients (age, educational status, social security, marital status), information about pregnancy (drugs used, status of their willingness to become pregnant, gestational week, status of attending examinations, status of collecting information about labour), the methods used to cope with the pain, and open-ended questions that evaluate the previous use of massage.
2. Birth Action Follow-Up Form: The questions that indicate the length of the first phase, the interventions performed to shorten the first phase of labour, the methods used by the patient to cope with the labour pain, the emotional behaviours of the pregnant women during labour, the length of the second phase, adjustment of the pregnant women, the presence of intervention in labour, the status of episiotomy, the total duration of labour and the baby's health.
3. Postpartum Interview Form: Open and closed questions that indicate the pregnant women's thoughts about labour, the status of overall satisfaction with labour and how the women feel were included in this form, which was prepared by a researcher in accordance with the relevant literature.
4. Visual Analogue Scale (VAS): The Visual Analogue Scale (VAS) was used to measure the severity of labour pain. On this scale, numbers from 0 to 10 appear on a horizontal line of 100 mm. The pain level is expressed in figures that range from 0 to 10, as follows: the absence of pain is indicated by "0", while the most severe pain is indicated by "10". In this method, it is explained to the individual that there are two endpoints and that he/she is free to mark any point that defines his/her pain.

   The VAS was applied to the participants in the control group three times in the latent (3-4 cm), active (5-7 cm) and transition phases (8-10 cm) of labour. The VAS was also applied to those in the experimental group two times before and after the massage in each phase. The diagnosis was made in accordance with the subjective data including the patient's verbal expression.
5. State-Trait Anxiety Inventory (STAI FORM TX-I): To determine state and trait anxiety levels of the participants, the state-trait anxiety inventory (STAI FORM TX -I) was used. The individual is required to indicate the feelings or behaviours that he/she has experienced in a specific situation according to the degree of severity by marking one of the options such as (1) Never, (2) Little, (3) Very and (4) Completely. The state-trait anxiety inventory requires the individual to describe how he/she feels at a certain moment and under certain conditions by considering his/her feelings about a specific situation. While high scores indicate high anxiety levels, low scores indicate low anxiety levels. The state-trait anxiety inventory consists of 20 statements. The score obtained from the scale may vary between 20 and 80. While a high score represents a high anxiety level, a low score represents a low anxiety level. In the scoring performed in accordance with the criteria directive, 0-19 points are regarded as "none", 20-39 points are regarded as "mild anxiety", 40-59 points are regarded as "moderate anxiety", 60-79 points are regarded as "heavy anxiety" and 80 points are regarded as "severe anxiety". In our study, the STAI FORM TX-I was used in the active (5-7 cm) phase in the control group and in the active (5-7 cm) phase after the massage in the experimental group to evaluate the anxiety experienced by women during labour.

Data Collection

After approval and permission to conduct the study were obtained from the ethics committee, the hospital's head nurse, delivery room charge nurse/midwife and other midwives and nurses were interviewed and informed about the purpose and scope of the study. Data were collected by one of the researchers. The researcher was aware of which patients were assigned to each group. However, the researchers did not interfere in any way with the study results. When they encountered women who met the inclusion criteria of the study, the purpose of the study was explained, and written consents were received from those who agreed to participate in the study. For the women who satisfied the criteria, participation in the study was voluntary. Additionally, during the study, no women requested to withdraw and no women were excluded from the study. Routine care and treatments for the women continued during data collection.

Procedure

Before the research data were collected, an informative meeting regarding the purpose and scope of the study was held for the members of the healthcare team who worked in the obstetrics and gynaecology clinic of the Turkish Republic Ministry of Health Public Hospitals Administration of Turkey, at the Istanbul Province xxx Training and Research Hospital, where the study would be conducted. In addition, cooperation was provided by the members of the healthcare team. For the correct application of the massage, the researcher was trained by the physical therapist who work at hospital. The massage was applied only to the pregnant women in the intervention group at every phase of labour. There was no intervention in the control group except for routine hospital applications. The steps taken in this study are discussed below.

For the pregnant women included in the experimental group:

* One-on-one interviews were conducted with the pregnant women, and the voluntary disclosure forms, which explained the purpose of the study, were completed.
* The prepared questionnaire form was applied.
* In addition to providing them with routine nursing/midwifery care, the women in the experimental group were administered a massage to the sacral region under the supervision of a doctor for 30 minutes using the effleurage (patting) ( 15 minutes) and vibration technique ( 15 minutes) in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour. To achieve this, the patients were placed in the left lateral position in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases of labour.
* The state-trait anxiety inventory (STAI FORM TX-I) was applied and evaluated after the massage in the active (5-7 cm) phase.
* The Visual Analogue Scale (VAS) was evaluated once after the massage in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases.
* Birth action follow-up form and postpartum interview forms were applied.

For the pregnant women included in the control group:

* One-on-one interviews were conducted with the pregnant women, and the voluntary disclosure forms, which explained the purpose of the study, were completed.
* The prepared questionnaire form was applied.
* Routine nursing/midwifery care was applied.
* The state-trait anxiety inventory (STAI FORM TX-I) was applied and evaluated in the active (5-7 cm) phase.
* The Visual Analogue Scale (VAS) was evaluated once in the latent (3-4 cm), active (5-7 cm) and transition (8-10 cm) phases.
* Birth action follow-up form and postpartum interview forms were applied One-on-one interviews were conducted with the women in both groups, and the voluntary disclosure forms, which explained the purpose of the study, were completed. After the prepared questionnaire form was applied to the women in the experimental group, routine nursing/midwifery care was provided.

Data analysis

In the evaluation of the data, in addition to descriptive statistical methods (e.g., percentage, frequency, mean, and standard deviation), the chi-square test and Student's t-test were used in the comparison of the qualitative data. The results were evaluated at a significance level of p <0.05.

The dependent variables of the study are the pain score averages of the pregnant women, the duration of the latent, active and transition phases of labour, and the anxiety level score. The independent variables of the study are the pregnant women's age, educational status, working status, and prenatal educational status, as well as the educational status of the husbands of the pregnant women, their willingness to become pregnant and the willingness to serve as controls before labour.

ELIGIBILITY:
Inclusion Criteria:

1. 19-40-year-old primiparous pregnant women;
2. Singleton pregnancies between 38-42 weeks;
3. Pregnant women whose labour began spontaneously;
4. Pregnant women with a healthy foetus;
5. Pregnant women without any complications that may cause dystocia during labour;
6. Pregnant women for whom analgesia and anaesthesia were not used during the first phase of labour;
7. Pregnant women who volunteered to participate in the research and who could establish verbal communication.

Exclusion Criteria:

1. Pregnant women with high-risk pregnancies, with caesarean section indication, and
2. Pregnant women with a chronic illness were excluded.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant woman
Enrollment: 60 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
The state-trait anxiety inventory (STAI FORM TX-I) evaluated | 6 hours
  The state-trait anxiety inventory (STAI FORM TX-I) was applied and evaluated after the massage in the active (5-7 cm) phase.To determine state and trait anxiety levels of the participants, the state-trait anxiety inventory (STAI FORM TX -I) was used. The individual is required to indicate the feelings or behaviours that he/she has experienced in a specific situation according to the degree of severity by marking one of the options such as (1) Never, (2) Little, (3) Very and (4) Completely.the STAI FORM TX-I was used in the active (5-7 cm) phase in the control group and in the active (5-7 cm) phase after the massage in the experimental group to evaluate the anxiety experienced by women during labour.

SECONDARY OUTCOMES:
The Visual Analogue Scale (VAS) evaluated | 6 hours
  The Visual Analogue Scale (VAS) was used to measure the severity of labour pain. On this scale, numbers from 0 to 10 appear on a horizontal line of 100 mm. The pain level is expressed in figures that range from 0 to 10, as follows: the absence of pain is indicated by "0", while the most severe pain is indicated by "10". In this method, it is explained to the individual that there are two endpoints and that he/she is free to mark any point that defines his/her pain.The VAS was applied to the participants in the control group once in the latent (3-4 cm), active (5-7 cm) and transition phases (8-10 cm) of labour. The VAS was also applied to those in the experimental group once after the massage in each phase.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Çevik, phD, Study Director — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mortazavi SH, Khaki S, Moradi R, Heidari K, Vasegh Rahimparvar SF. Effects of massage therapy and presence of attendant on pain, anxiety and satisfaction during labor. Arch Gynecol Obstet. 2012 Jul;286(1):19-23. doi: 10.1007/s00404-012-2227-4. Epub 2012 Jan 21. PMID 22271239
- [Result] Abbaspoor, Z., Mohammadkhani, S.L. (2013). Lavender aromatherapy massages in reducing labor pain and duration of labor: A randomized controlled trial. African Journal of Pharmacy and Pharmacology, 7(8): 426-430. DOI: 10.5897/AJPP12.391.
- [Result] Fenwick J, Staff L, Gamble J, Creedy DK, Bayes S. Why do women request caesarean section in a normal, healthy first pregnancy? Midwifery. 2010 Aug;26(4):394-400. doi: 10.1016/j.midw.2008.10.011. Epub 2008 Dec 30. PMID 19117644
- [Result] Field T. Pregnancy and labor massage. Expert Rev Obstet Gynecol. 2010 Mar;5(2):177-181. doi: 10.1586/eog.10.12. PMID 20479957
- [Result] Silva Gallo RB, Santana LS, Jorge Ferreira CH, Marcolin AC, Polineto OB, Duarte G, Quintana SM. Massage reduced severity of pain during labour: a randomised trial. J Physiother. 2013 Jun;59(2):109-16. doi: 10.1016/S1836-9553(13)70163-2. PMID 23663796
- [Result] Bolbol-Haghighi N, Masoumi SZ, Kazemi F. Effect of Massage Therapy on Duration of Labour: A Randomized Controlled Trial. J Clin Diagn Res. 2016 Apr;10(4):QC12-5. doi: 10.7860/JCDR/2016/17447.7688. Epub 2016 Apr 1. PMID 27190898
- [Result] Hosseini SE, Bagheri M, Honarparvaran N. Investigating the effect of music on labor pain and progress in the active stage of first labor. Eur Rev Med Pharmacol Sci. 2013 Jun;17(11):1479-87. PMID 23894767
- [Result] Janssen P, Shroff F, Jaspar P. Massage therapy and labor outcomes: a randomized controlled trial. Int J Ther Massage Bodywork. 2012;5(4):15-20. doi: 10.3822/ijtmb.v5i4.164. Epub 2012 Dec 19. PMID 23429706
- [Result] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342

DOCUMENTS (3):
  • Statistical Analysis Plan: statistical analysis (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03755284/SAP_000.pdf
  • Informed Consent Form: Informed Consent Form (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03755284/ICF_001.pdf
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03755284/Prot_002.pdf